CLINICAL TRIAL: NCT07316998
Title: Incidence of Myopia in a Prospective Cohort of Emmetropic Children and Associated Ocular and Environmental Factors
Acronym: PREMYOP
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: TCN_2025_8
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 4 to 8 years at inclusion, emmetropic (cycloplegic SE 0 to +2D) in each eye d
  Interventions: Other: annual follow-up

INTERVENTIONS:
Other: annual follow-up — annual follow-up including ophtalmologic examination and biometry and behavioural questionnaires

SUMMARY:
Myopia and high myopia are among the leading causes of visual impairment and blindness worldwide. The total number of people with myopia worldwide was estimated at 2.6 billion in 2020 and could reach 4.8 billion by 2050 unless preventive interventions are implemented.

Most epidemiological studies have focused on risk factors for myopia progression, with far fewer addressing the factors that cause a child to shift from emmetropia to myopia. The risk factors for the onset of myopia may be the same as those for myopia progression. However, for an equivalent level of risk exposure, it remains unclear why some children develop myopia while others do not.

Identifying the population most at risk of developing myopia would make it possible to propose preventive treatments aimed at delaying or preventing its onset. This would allow evaluation of the effectiveness of current myopia control treatments (peripheral defocus lenses, atropine, contact lenses) in preventing the onset of myopia, as well as future targeted treatments, including the potential benefit of early optical correction-a strategy once used but later abandoned due to a lack of robust scientific evidence.

The establishment of longitudinal follow-up of young emmetropic children at the French Institute of Myopia will enable the acquisition of high-quality imaging, allowing investigation of the association between advanced imaging parameters and external environmental factors with the onset of myopia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years and < 9 years
* Spherical equivalent measured by autorefractometer ≥ 0.00 and ≤ +2.00 diopters in each eye (cycloplegic autorefraction)

Exclusion Criteria:

* Presence of trauma in at least one eye
* Presence of inflammatory ocular pathology in at least one eye
* History of intraocular pressure-lowering ophthalmic treatment, intravitreal injections, laser treatment, or myopia control therapy (e.g., atropine, orthokeratology, myopia control lenses)
* History of ophthalmic surgery other than for the management of strabismus (e.g., cataract surgery, filtering surgery, intravitreal surgery) in at least one eye

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 4 to 8 years at inclusion, emmetropic (cycloplegic refractive error between 0 and +2 diopters - inclusive - in spherical equivalent in each eye).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
To describe the incidence of myopia over the 2 years following inclusion in emmetropic children. | Annual follow up : Year 1 and year 2
  Onset of myopia within the 2 years following inclusion, defined as a spherical equivalent (SE) ≤ -0.50 D in at least one eye. Measurement of the spherical equivalent will be performed under cycloplegia using an autorefractor.

SECONDARY OUTCOMES:
To describe the incidence of myopia over the 5 years following inclusion in emmetropic children. | annual follow-up until Year 5
  Onset of myopia within the 5 years following inclusion, defined as a spherical equivalent (SE) ≤ -0.50 D in at least one eye. Measurement of the spherical equivalent will be performed under cycloplegia using an autorefractor.